CLINICAL TRIAL: NCT00427583
Title: An Open-label Multicenter Phase II Study of Imatinib Mesylate Treatment of Patients With Malignant Peripheral Nerve Sheath Tumors
Brief Title: Imatinib Mesylate Treatment of Patients With Malignant Peripheral Nerve Sheath Tumors
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: stopped due to slow recruitment and no effect
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE57
Record Dates: First submitted 2007-01-25; First posted 2007-01-29 (Estimated); Last update posted 2012-08-07 (Estimated); Status verified 2012-08

CONDITIONS: Malignant Peripheral Nerve Sheath Tumors
Keywords: Malignant,; peripheral,; nerve sheath tumors,; MPNST,; neurofibromatosis,; NF1,; Imatinib mesylate
MeSH Terms: conditions — Neurofibrosarcoma; Nerve Sheath Neoplasms; Neurofibromatoses | interventions — Imatinib Mesylate

ARMS (1):
- STI571 (Experimental)
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
This study assesses the safety and efficacy of imatinib mesylate treatment of patients with malignant peripheral nerve sheath tumors

ELIGIBILITY:
Inclusion criteria:

* Patients ≥18 years of age
* Histologically documented diagnosis of malignant MPNST
* Unresectable local MPNST or metastatic MPNST and therefore incurable with any conventional multimodality approach Life expectancy of at least 6 months.

Exclusion criteria:

* Patient has received any other investigational agents within 28 days of first day of study drug dosing.
* Chemotherapy and or radiotherapy in between the last 6 weeks before study entry, surgery in between the last 14 days before study entry.
* Female patients who are pregnant or breast feeding or women of child bearing potential who are not using a highly effective method of birth control.
* Known CNS metastases

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Response rate assessed by a Tumor MRI scan every 6 weeks or if clinically indicated. | Every 36 weeks

SECONDARY OUTCOMES:
Time to progression assessed by an MRI scan. | Every 36 weeks
Overall survival | Every 36 weeks
Safety and tolerability assessed by abnormal lab values (hematology, biochemistry, urinalysis), by physical examination and vital signs | Every 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (2):
- Germany (2):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Hamburg